CLINICAL TRIAL: NCT02251132
Title: An Open-label, Parallel Group, Multiple-dose Investigation of the Pharmacokinetics of Tipranavir Soft Elastic Capsules SEDDS and Ritonavir Soft Gel Capsules and Their Effects on Cytochrome P-450 (3A4) Activity in Normal Healthy Volunteers
Brief Title: Pharmacokinetics of Tipranavir Soft Elastic Capsules (SEDDS) and Ritonavir and Their Effects on Cytochrome P-450 (3A4) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1182.5
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Healthy

ARMS (8):
- TPV/RTV Low 1 (Experimental)
  Interventions: Drug: TPV low 1; Drug: Ritonavir high; Drug: Radiolabelled erythromycin
- TPV/RTV Low 2 (Experimental)
  Interventions: Drug: TPV low 2; Drug: RTV low; Drug: Radiolabelled erythromycin
- TPV/RTV Low 3 (Experimental)
  Interventions: Drug: TPV low 2; Drug: Ritonavir high; Drug: Radiolabelled erythromycin
- TPV/RTV Medium 1 (Experimental)
  Interventions: Drug: TPV medium; Drug: RTV low; Drug: Radiolabelled erythromycin
- TPV/RTV Medium 2 (Experimental)
  Interventions: Drug: TPV medium; Drug: Ritonavir high; Drug: Radiolabelled erythromycin
- TPV/RTV High 1 (Experimental)
  Interventions: Drug: TPV high 1; Drug: RTV low; Drug: Radiolabelled erythromycin
- TPV/RTV High 2 (Experimental)
  Interventions: Drug: TPV high 1; Drug: Ritonavir high; Drug: Radiolabelled erythromycin
- TPV/RTV High 3 (Experimental)
  Interventions: Drug: TPV high 2; Drug: Ritonavir high; Drug: Radiolabelled erythromycin

INTERVENTIONS:
Drug: TPV low 1
  Arms: TPV/RTV Low 1
Drug: TPV low 2
  Arms: TPV/RTV Low 2; TPV/RTV Low 3
Drug: TPV medium
  Arms: TPV/RTV Medium 1; TPV/RTV Medium 2
Drug: TPV high 1
  Arms: TPV/RTV High 1; TPV/RTV High 2
Drug: TPV high 2
  Arms: TPV/RTV High 3
Drug: RTV low
  Arms: TPV/RTV High 1; TPV/RTV Low 2; TPV/RTV Medium 1
Drug: Ritonavir high
  Arms: TPV/RTV High 2; TPV/RTV High 3; TPV/RTV Low 1; TPV/RTV Low 3; TPV/RTV Medium 2
Drug: Radiolabelled erythromycin

SUMMARY:
The objective of this study is to establish the tipranavir-ritonavir steady-state dose-exposure relationships when administered on a b.i.d. dosing regimen; to determine the effects of tipranavir (TPV) and ritonavir (RTV) on cytochrome P-450 (CYP3A4) activity; to establish the dependency of the TPV M1 metabolite on RTV co-administration. Additionally, the short-term safety and tolerance of this drug combination will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 75 years of age inclusive
* Female subjects of child-bearing potential are required to use a barrier contraceptive method for at least 3 months prior to administration of study medication, during study medication administration and for 30 days after the end of the study
* Ability to swallow numerous large capsules without difficulty
* A body mass index (BMI) between 19 and 29 kg/m2
* Signed informed consent prior to trial participation
* Reasonable probability for completion of the study
* Acceptable screening laboratory values that indicate adequate baseline organ function are required at the time of screening. Laboratory values are considered to be acceptable if severity is no higher than Grade 1 based on the AIDS Clinical Trials Group (ACTG) Grading Scale. All laboratory values > Grade 1 are subject to approval by the BIPI clinical monitor
* Acceptable medical history, physical examination, electrocardiogram, and chest X-ray are required prior to entering the treatment phase of the study
* Willingness to abstain from alcohol for 48 hours prior to study Day 0 and abstain from alcohol for the duration of the study
* Willingness to abstain from ingesting grapefruit or grapefruit juice for the duration of the study
* Urine drug screen negative for drugs of abuse
* Negative HIV serology
* Negative for Hepatitis B surface antigen and Hepatitis C antibody

Exclusion Criteria:

* Female subjects who:

  * have a positive serum pregnancy test at Visits 1 or 2 OR
  * are breastfeeding
* Receipt of any other investigational medicine for 30 days prior to Day 0
* Receipt of any known enzyme altering drug for 30 days prior to Day 0, grapefruit and grapefruit juice within 15 days prior to Day 0 and antibiotics within 10 days prior to Day 0
* Excessive cigarette smoking, defined as greater than 10 cigarettes per day
* Blood or plasma donation within 30 days prior to Day 0
* Subjects with a seated systolic blood pressure either < 100 mg Hg or > 150 mm Hg; resting heart rate either < 50 beats/min or > 90 beats/min
* Subjects with a history of any illness or allergy that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering tipranavir or ritonavir to the subject
* Subjects who have had an acute illness within 2 weeks prior to Day 0
* Subjects who are currently taking any over-the-counter drug within 7 days prior to Day 0, or who are currently taking any prescription drug that, in the opinion of the investigator in consultation with the BIPI medical monitor and pharmacokineticist, might interfere with either the absorption, distribution or metabolism of the test substances
* Hypersensitivity to tipranavir, ritonavir or sulfonamide containing drugs
* Evidence of active substance abuse that, in the investigator's opinion, could affect study adherence

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2000-10; Primary Completion 2000-12 (Actual)

PRIMARY OUTCOMES:
Trough plasma concentration at steady state (Cmin,ss) | up to 24 hours
Maximum plasma concentration at steady state (Cmax,ss) | up to 24 hours
Time of maximum concentration (tmax) | up to 24 hours
Area under the plasma concentration time curve from 0 to 12 hours (AUC0-12) | up to 12 hours

SECONDARY OUTCOMES:
Oral clearance (Cl/F) | up to 24 hours
Apparent terminal half life (t1/2) | up to 24 hours
Percent of erythromycin metabolized per hour | up to 24 hours
  Erythromycin breath test (ERMBT)
Number of subjects with clinically significant findings in laboratory tests | up to 32 days
Number of subjects with adverse events | up to 32 days